CLINICAL TRIAL: NCT04348032
Title: Apatinib Combined With PLD vs PLD for Platinum-resistant Recurrent Ovarian Cancer(APPROVE): a Randomized, Controlled, Open-label, Phase 2 Trial
Brief Title: Apatinib Combined With PLD vs PLD for Platinum-resistant Recurrent Ovarian Cancer
Acronym: APPROVE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ling-Ying Wu, chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016YFC1303704
Record Dates: First submitted 2020-04-14; First posted 2020-04-15 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Platinum-resistant Recurrent Ovarian Cancer
MeSH Terms: interventions — 1-dodecylpyridoxal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLD (Active Comparator): PLD 40 mg/m2 D1 ivgtt q4w
  Interventions: Drug: PLD 40mg/m2 ivgtt q4w
- PLD + Apatinib (Experimental): PLD 40 mg/m2 D1 ivgtt q4w + Apatinib 250mg po qd
  Interventions: Drug: PLD 40mg/m2 ivgtt q4w +Apatinib 250mg po qd

INTERVENTIONS:
Drug: PLD 40mg/m2 ivgtt q4w +Apatinib 250mg po qd — Patients receive PLD and apatinib at the same time. The dose of intravenous chemotherapy drug is calculated according to the body surface area, and the dose of oral drug apatinib is 250mg qd. Dose suspension and dose reduction are allowed only when patients have serious adverse reactions. The intravenous chemotherapy drug PLD dose is only allowed to be down-regulated twice (one time is to reduce the standard dose by 25%), and the oral drug apatinib dose is only allowed to be reduced once (250mg gravity QD changed to 250mg gravity Qod). Otherwise the patients will drop out of the study.
  Arms: PLD + Apatinib
Drug: PLD 40mg/m2 ivgtt q4w — The dose of intravenous chemotherapy drug is calculated according to the body surface area. When patients have serious adverse reactions, dose suspension and dose reduction are allowed. The PLD dose is only allowed to be down-regulated twice (one time is to reduce the standard dose by 25%).
  Arms: PLD

SUMMARY:
Epithelial ovarian cancer is the most fatal gynecological malignancy. Despite initial therapeutic response, the majority of advanced-stage patients relapse and eventually succumb to chemoresistant disease. The prognosis of patients with platinum-resistant or refractory ovarian cancer was very poor, with the response rate of 20%~25% after chemotherapy. The purpose of treatment for recurrent ovarian cancer is mainly to improve the quality of life of patients and prolong survival. Angiogenesis is essential for tumor growth and metastasis.And VEGF/VEGF receptor(VEGFR) signaling pathway is the most promising angiogenic target due to its key roles in angiogenesis and tumor growth.This study sought to assess the efficacy and safety of the combination therapy of apatinib and PLD, clarifying whether combination therapy could improve the outcomes of patients with platinum-resistant recurrent ovarian cancer.

DETAILED DESCRIPTION:
This study is a randomized, parallel-controlled, multicenter clinical study. We recruit patients over the age of 18 years with platinum-resistant recurrent ovarian cancer. patients who meet the criteria for enrollment are randomly divided into two groups, including experiment group and control group. This study will be divided into three stages: 1. Baseline period (within 21 days before the start of treatment): Patients will complete screening tests during the baseline period to assess whether they meet the selection criteria. 2. Treatment period (from the first administration to the completion of the last treatment cycle). The tumor will be evaluated every 8 weeks during this period. If the treatment is effective, the chemotherapy does not exceed 6 cycles，then experiment group receives oral apatinib maintenance therapy until the disease progresses or toxicity could not be tolerated. Control group is followed up. 3. Follow-up period. After the end of chemotherapy, the survival status and follow-up anti-tumor therapy are collected by telephone or research centers visit every 3 months until death or loss of follow-up.The primary endpoint is the progression-free survival time(PFS) of patients and is judged according to Response Evaluation Criteria in Solid Tumors, version 1.1. Adverse events are classified and recorded according to the National Cancer Institute's Standard of Common terms for adverse reactions (NCI-CTCAE) version 4.0.

ELIGIBILITY:
Inclusion criteria

1. Patients were diagnosed with ovarian cancer, fallopian tube cancer or primary peritoneal cancer confirmed by previous pathology, and the pathological type was non-mucinous adenocarcinoma.There were previous surgical wax preservation.
2. Initial platinum-resistant relapse, the recurrence time was less than 6 months after the last chemotherapy.
3. Complicated with malignant pleural effusion or ascites, or with recurrent lesions that can be evaluated clinically.
4. ECOG physical status score 0 or 1.
5. The expected survival time is ≥ 4 months.
6. In the previous treatment, there was no antivascular targeted therapy;
7. Patients without pleural effusion or ascites should be confirmed by CT or MRI according to the standard of RECIST1.1 version, requiring the patient to have at least one measurable focus as the target focus. If the target focus is a lymph node with a short diameter of more than 1.5 cm, and the target focus is not suitable for surgical treatment, the target focus has not received radiotherapy or relapsed in the radiotherapy field.
8. The baseline blood routine conforms to the following criteria:

   1. neutrophil count ≥ 1.5x109 /L;
   2. platelet count ≥ 100x109 PG L;
   3. hemoglobin ≥ 9g/dL (blood transfusion is allowed to achieve or maintain this target) .
9. Liver function meets the following criteria:

   1. total bilirubin<1.5 normal limit (ULN);
   2. glutamic oxaloacetic transaminase (AST), glutamic pyruvic transaminase (ALT)<2.5xULN, which is allowed<5xULN in patients with liver metastasis.
10. Serum creatinine ≤ 1.25xULN or calculated creatinine clearance ≥ 50mL/min.

Exclusion criteria

1. Have received more than two chemotherapy regimens in the past.
2. Currently or recently (within 30 days before enrollment) using another research drug or participating in another clinical study.
3. other malignant tumors have occurred within 5 years (except adequately treated cervical carcinoma in situ or skin squamous cell carcinoma, or controlled basal cell carcinoma of the skin).
4. Patients with hypertension that cannot be reduced to normal range after antihypertensive treatment (systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥ 90 mmHg).
5. Suffer from myocardial ischemia or myocardial infarction above II grade and poorly controlled arrhythmias (including QTc interval ≥ 470ms in females).
6. According to the NYHA standard, there were previous or present cardiac insufficiency of grade II or above, or color Doppler echocardiography showed that the left ventricular ejection fraction ((LVEF)) was less than 50% or the lower limit of the normal value.
7. Abnormal coagulation function (INR>1.5 or prothrombin time (PT) > ULN+4 seconds or APTT>1.5xULN), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy.
8. There were significant clinical bleeding symptoms or definite bleeding tendency in the first 3 months, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood or above, or suffering from vasculitis.
9. Major surgical operations or severe traumatic injuries, fractures or ulcers occurred within the first 4 weeks of randomization.
10. There are significant factors affecting oral drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction.
11. Urine routine indicates urinary protein ≥++, or confirms 24-hour urinary protein ≥ 1.0g.
12. The researchers judged other conditions that may affect the conduct of clinical studies and the determination of research results.
13. Allergic or heterogeneous reactions to doxorubicin and / or related substances.
14. The cumulative dose of doxorubicin (including previous anthracycline, if any) is expected to reach or exceed 550 mg after 4 courses of doxorubicin liposome injection treatment.
15. Uncontrollable arrhythmias or electrocardiograms abnormalities determined by the lead researcher to be at risk.
16. A history of doxorubicin liposome therapy in recent half a year.
17. Have previously received local radiotherapy of the pelvis or lower abdomen.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival(PFS) | up to 2 years
  From date of randomization until the date of first documented progression or died

SECONDARY OUTCOMES:
Overall survival(OS) | up to 2 years
  From date of randomization until the date of death from any cause
Objective response rate(ORR) | up to 2 years
  The proportion of patients with tumor shrinkage reaching a certain amount and for a certain period of time, including cases of CR PR.
disease control rate(DCR) | up to 2 years
  including CR, PR, SD
hematological toxicity and non-hematological toxicity | up to 2 years
  including hematological toxicity and non-hematological toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, MD, Study Chair — Chinese Academy of Medical Sciences
Locations (16):
- China (16):
  - National Cancer Center/ National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Beijing Obstetrics and Gynecology Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Guangxi Cancer Hospital, Guangxi, Guangxi
  - Hubei Cancer Hospital, Hubei, Hubei
  - Hunan Cancer Hospital, Hunan, Hunan
  - Xiangya Hospital of Central South University, Hunan, Hunan
  - The first Hospital of Jilin University, Jilin, Jilin
  - Liaoning Cancer Hospital, Liaoyang, Liaoning
  - Shandong Cancer Hospital, Shangdong, Shangdong
  - Tumor Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Tumor Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Yunnan, Yunnan

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Wang T, Tang J, Yang H, Yin R, Zhang J, Zhou Q, Liu Z, Cao L, Li L, Huang Y, Jiang K, Wang W, She F, Guan N, Hou Z, Li N, Wu L. Effect of Apatinib Plus Pegylated Liposomal Doxorubicin vs Pegylated Liposomal Doxorubicin Alone on Platinum-Resistant Recurrent Ovarian Cancer: The APPROVE Randomized Clinical Trial. JAMA Oncol. 2022 Aug 1;8(8):1169-1176. doi: 10.1001/jamaoncol.2022.2253. PMID 35771546